CLINICAL TRIAL: NCT04699214
Title: A Prospective, Randomized Controlled Phase II Clinical Study Evaluating the Efficacy and Safety of Endostar Combined With AI Regimen Compared With AI Regimen in Adjuvant Treatment After Radical Resection of Recurrent Soft Tissue Sarcoma
Brief Title: Endostar Combined With AI Regimen Compared With AI in Adjuvant Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Chen (Other)
Responsible Party: Sponsor-Investigator, Yong Chen, Chief Physician, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1906203-3
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Other Disorders of Soft Tissues
Keywords: OS（Overall Survival）; EFS（Event-Free Survival Rate）
MeSH Terms: interventions — endostar protein; Endostatins

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled, open phase II clinical study
Who Masked: Participant
Masking Description: The dose of Endostar is not adjusted, and the specific adjustment plan of the chemotherapy regimen is adjusted according to the clinical experience of the investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endostar combined with chemotherapy AI (Experimental): Endostar: Endostar 45mg/d, D1-5 iv, Q3W, that is, continuous intravenous pump injection for 120 hours for 5 consecutive days, one cycle. Endostar uses 15 medicines per cycle, 15 Endostar medicines and a Baxter pump per single cycle. Subjects buy and use them at their own expense every two cycles.
  AI: Doxorubicin (ADM) 60mg/m2 iv D1+ Ifosfamide (IFO) 2g/m2/d D1-5+ Mesna 400mg/m 2 (ifosfamide start infusion, time after infusion 4 hours, 8 hours injection) D1-5, Q3W.
  Interventions: Drug: Endostar (recombinant human endostatin injection)
- Chemotherapy AI (Active Comparator): AI: Doxorubicin (ADM) 60mg/m2 iv D1+ Ifosfamide (IFO) 2g/m2/d D1-5+ Mesna 400mg/m 2 (ifosfamide start infusion, time after infusion 4 hours, 8 hours injection) D1-5, Q3W.
  Interventions: Drug: Chemotherapy AI
- Observation group (Placebo Comparator): The dose of Endostar is not adjusted, and the specific adjustment plan of the chemotherapy regimen is adjusted according to the clinical experience of the investigator.
  Patients with no disease progression (local tumor recurrence, distant metastasis, or the appearance of new lesions of the same tumor subtype) and the adverse reactions can be tolerated, continue to use the drug for 6 cycles, and cannot receive other anti-tumor treatments. In the course of medication, if the disease progresses or the researcher believes that the patient is not suitable for continuing medication, the medication will end.
  Interventions: Drug: Endostar (recombinant human endostatin injection)

INTERVENTIONS:
Drug: Endostar (recombinant human endostatin injection) — The experimental group is Endostar combined with AI
  Arms: Endostar combined with chemotherapy AI; Observation group
Drug: Chemotherapy AI — AI: Doxorubicin (ADM) 60mg/m2 iv D1+ Ifosfamide (IFO) 2g/m2/d D1-5+ Mesna 400mg/m 2 (ifosfamide start infusion, time after infusion 4 hours, 8 hours injection) D1-5, Q3W
  Arms: Chemotherapy AI

SUMMARY:
To evaluate the effectiveness, safety and tolerability of Endostar (recombinant human endostatin) combined with AI chemotherapy in adjuvant treatment after radical resection of recurrent soft tissue sarcoma.

DETAILED DESCRIPTION:
Eligible patients with stage IIB/III soft tissue sarcoma after surgical treatment for local recurrence were randomly divided into three groups:

Group A: Endostar combined chemotherapy AI Endostar: Endostar 45mg/d, D1-5 iv, Q3W, that is, continuous intravenous pump injection for 120 hours for 5 consecutive days, one cycle. Endostar takes 15 medicines per cycle, and a Baxter pump per single cycle. Subjects buy and use them at their own expense every two cycles.

AI: Doxorubicin (ADM) 60mg/m2 iv D1+ Ifosfamide (IFO) 2g/m2/d D1-5+ Mesna 400mg/m 2 (ifosfamide start infusion, time after infusion 4 hours, 8 hours injection) D1-5, Q3W.

Group B:Chemotherapy AI AI: Doxorubicin (ADM) 60mg/m2 iv D1+ Ifosfamide (IFO) 2g/m2/d D1-5+ Mesna 400mg/m 2 (ifosfamide start infusion, time after infusion 4 hours, 8 hours injection) D1-5, Q3W.

Group C: Observation group Best supportive treatment, observation and follow-up. The dose of Endostar is not adjusted, and the specific adjustment plan of the chemotherapy regimen is adjusted according to the clinical experience of the investigator.

Patients with no disease progression (local tumor recurrence, distant metastasis, or the appearance of new lesions of the same tumor subtype) and the adverse reactions can be tolerated, continue to use the drug for 6 cycles, and cannot receive other anti-tumor treatments. During the medication, if the disease progresses or the researcher believes that the patient is not suitable for continuing medication, the medication will end.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with soft tissue sarcoma confirmed by histopathology and cytology;
2. Patients with soft tissue sarcoma judged to be stage IIB/III according to the AJCC staging of soft tissue sarcoma;
3. Patients who have previously undergone surgery can be included in the group, but according to the researcher's evaluation, they must have recovered and the operation completion time is at least 4 weeks from the study entry;
4. Local radiotherapy can be received during chemotherapy;
5. Have received anti-tumor drug treatment in the past, including adjuvant or neoadjuvant chemotherapy, but it has been over 6 months before the start of the study treatment;
6. R0 resection after local recurrence, non-chemotherapeutic resistant soft tissue sarcoma, including synovial sarcoma, pleomorphic liposarcoma, myxoid/round cell liposarcoma, pleomorphic undifferentiated sarcoma, leiomyosarcoma, myxofibrosarcoma, Angiosarcoma, malignant peripheral nerve sheath tumor, epithelioid sarcoma, etc., except Ewing's sarcoma, embryonic/acinoid rhabdomyosarcoma and other sarcomas that do not use AI regimen as the first-line chemotherapy regimen, and some chemotherapy-insensitive sarcomas: highly differentiated/removed Differentiated liposarcoma, clear cell sarcoma, alveolar soft tissue sarcoma, extraosseous mucinous chondrosarcoma, etc.;
7. No gender limit, ≥18 years old;
8. ECOG score ≤ 2;
9. The expected survival period is ≥3 months;
10. Sufficient blood function: absolute neutrophil count (ANC)≥1.5×109/L and platelet count≥80×109/L and hemoglobin≥9 g/dL;
11. Sufficient liver function: total bilirubin ≤ upper limit of normal (ULN); AST and ALT ≤ 1.5 times upper limit of normal (ULN); alkaline phosphatase ≤ 5 times upper limit of normal (ULN);
12. Sufficient renal function: serum creatinine ≤ upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min;
13. The electrocardiogram is basically normal, and there is no unhealed wound on the body;
14. Those who have not had a severe allergic reaction to biological agents, especially E. coli genetic engineering products;
15. Women of childbearing age must agree to use contraceptive measures (such as intrauterine device (IUD), contraceptives or condoms) during the study period and within 6 months after the end of the study; serum or urine pregnancy within 7 days before study entry The test is negative and must be a non-lactating patient; men should agree to use contraception during the study period and within 6 months after the end of the study period.
16. The patient voluntarily joined the study, signed an informed consent form, had good compliance, and was able to be followed up by the trial staff.

Exclusion Criteria:

1. Pregnant or lactating women, or female patients who are fertile but have not taken contraceptive measures;
2. There are severe acute infections that have not been controlled; or there are purulent and chronic infections, and the wounds do not heal;
3. There is a second primary tumor (except skin basal cell carcinoma);
4. Those who have participated in other drug clinical trials within 4 weeks.
5. Pre-existing severe heart disease, including: congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina, myocardial infarction, severe heart valve disease, and refractory hypertension;
6. People with uncontrollable neurological or mental illnesses or mental disorders, poor compliance, and unable to cooperate and describe the treatment response; primary brain tumors or central nerve metastases have not been controlled, and have obvious intracranial hypertension or neuropsychiatry Symptoms;
7. Those with bleeding tendency;
8. Evidence of hereditary hemorrhagic constitution or coagulopathy;
9. A clear history of allergy to chemotherapy drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
EFS （Event-Free Survival Rate） | 2 year
  Prospective observation of the 2-year event-free survival rate EFS (Event-Free Survival Rate) of recombinant human endostatin injection (Endostar, trade name: Endostar) combined with adjuvant chemotherapy for local recurrence of soft tissue sarcoma, ie no progress , No disease-related deaths, no time for new lesions.

SECONDARY OUTCOMES:
OS（Overall Survival） | 2 year
  To evaluate the OS (Overall Survival)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be announced after the clinical trial is over.